CLINICAL TRIAL: NCT05515653
Title: Impact of the Genetic Background as a Risk Factor for Atherosclerotic Cardiovascular Disease in the Brazilian Population
Acronym: CV-GENES
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Collaborators: Grupo Fleury (Unknown); Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Álvaro Avezum Junior, Principal Investigator, Hospital Alemão Oswaldo Cruz
Other Study IDs: HAlemaoOswaldoCruz; CAAE: 56482922.2.1001.0070 (Other: Brazilian National Ethics Committee)
Record Dates: First submitted 2022-08-01; First posted 2022-08-25 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Acute MI; Stroke; Peripheral Arterial Disease; Genetic Predisposition to Disease
Keywords: case-control study; Polymorphism genetic; cardiovascular disease; observational study
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Peripheral Arterial Disease; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total blood, Buffy Coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case - atherosclerotic cardiovascular disease: Patients with the first atherosclerotic cardiovascular event (Acute Myocardial Infarction, Stroke and Peripheral Artery Thrombotic-Ischemic Events)
  Interventions: Genetic: Exposure to genetics (polygenic)
- Control - without atherosclerotic cardiovascular disease ou healthy: Patients who sought medical care at the same site as cases without atherosclerotic cardiovascular event (Acute Myocardial Infarction, Stroke and Peripheral Artery Thrombotic-Ischemic Events) or healthy individuals
  Interventions: Genetic: Exposure to genetics (polygenic)

INTERVENTIONS:
Genetic: Exposure to genetics (polygenic) — The polygenic risk score (PRS) aggregates the effects of genetic variants into a single number that predicts the genetic predisposition to a phenotype. PRS are typically composed of hundreds to millions of genetic variants, usually Single Nucleotide Polymorphisms (SNPs). For each individual, the number of risk alleles computed in each variant is summed and weighted by the estimated value of the obtained effects (log odds ratio for traits with binary values or Beta coefficients for traits with continuous value) obtained from large-scale genomic studies ( GWAS)
  Other Names: polygenic risk score

SUMMARY:
The main objective of this project is to evaluate the genomic information previously associated with cardiovascular diseases (CVD) and its importance as an independent risk predictor (expressed in Odds Ratio) when adjusted for traditional risk factors (smoking, diabetes, arterial hypertension, obesity , anxiety and depression, inadequate diet, physical inactivity, alcohol consumption and apolipoprotein B/A1 ratio (ApoB/ApoA1).

An unpaired case-control study of individuals over 18 years of age will be carried out. Cases (N = 1867) will be enrolled right after the occurrence of the first atherosclerotic cardiovascular event (Acute Myocardial Infarction, Stroke and Peripheral Artery Thrombotic-Ischemic Events). The ratio between cases and controls will be 1:1. The controls (N = 1867) will be adult individuals over 18 years of age who sought medical care at the same locations for other clinical reasons (no CVD) or individuals without any overt disease. The genetic evaluation will be performed through the association of Low-covering Whole Genome Sequencing (coverage 0.5-5x) and Whole Exome Sequencing (average coverage 30x).

DETAILED DESCRIPTION:
The study will be carried out in about 50 centers, comprising the five Brazilian regions. The study will be conducted from July 2022 to December 2023. Data collection will be performed at each center consecutively, for cases and controls, through electronic Case Report Form (CRF).

Cases (N = 1867) will be selected by the occurrence of the first atherosclerotic cardiovascular event (Acute Myocardial Infarction, Stroke and Peripheral Arterial Thrombotic-Ischemic Events) during the hospitalization phase for the management of the acute atherothrombotic event. The ratio between cases and controls will be 1:1. Controls (N = 1867) will be adult individuals over 18 years of age who sought medical care at the same locations for other clinical reasons (no CVD) or individuals without any overt disease. The definitions of acute atherothrombotic events follow classic clinical and complementary exam criteria and are based on national and international guidelines. The complete project was submitted to the local Institutional Review Board (IRB)/National Research Ethics Commission (CONEP) system and has ethical approval (CAAE: 56482922.2.1001.0070). All cases and controls will be invited to participate and, if they agree, an Informed Consent Form will be obtained.

Investigators will assess exposures to traditional risk factors in combination with genomic data (polygenic risk score) in both cases and controls, and these exposures will be expressed as odds ratios. Multiple logistic regression models will be built to adjust and determine the strengths of association between demographic variables, traditional risk factors and genetic data: gender, age, ethnicity, weight, body mass index, smoking, diabetes, hypertension, obesity, anxiety and depression, inadequate diet, physical inactivity, alcohol consumption and apolipoprotein B/A1 ratio (ApoB/ApoA1). For each association variable with a greater chance of cardiovascular disease (significant OR), an attributable risk will be calculated to estimate the fraction of risk attributable to the genetic component (Polygenic Risk Score) and to other clinical and demographic variables.

The polygenic risk score will be calculated through a hybrid approach by taking into account the following features: effect size of each Single Nucleotide Polymorphism (SNP), number of effect alleles observed, sample ploidy, total number of SNPs included in the Polygenic Risk Score, and the number of nonmissing SNPs in the sample. Each risk allele will be given points in the risk score, and the total score will range between 0 (absence of risk alleles) and the maximum value (yet to be defined), based on the distribution of risk alleles that will be identified in the population included in the study. The scale will be interpreted in a direct (positive) association, i.e., the higher the score, the higher the number of alleles and respective weighted effect sizes. Finally, the polygenic risk score will be adjusted to previously reported traditional risk factors for atherosclerotic cardiovascular disease to determine the attributable risk fraction associated with the genomic profile.

ELIGIBILITY:
Inclusion Criteria:

* Cases: adults over 18 years with first atherosclerotic cardiovascular event (Acute Myocardial Infarction, Stroke and Peripheral Artery Thrombotic-Ischemic Events)
* Controls: adult individuals over 18 years of age who sought medical care at the same locations for other clinical reasons (no CVD) or individuals without any overt disease

Exclusion Criteria:

* Previous occurrence of Cardiovascular Event (Myocardial Infarction, Stroke or Peripheral Artery Thrombotic Events
* Patients already recruited in another study linked to the GENOMA Brazil Program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In-hospital patients with the first atherosclerotic event will be enrolled (Cases). Patients being attended in the same hospitals without cardiovascular events or without any overt disease will be the controls. The sample size calculation assumed a dominant inheritance pattern, within a non-matched case-control study design 1:1. A sample of 1867 cases and 1867 controls would have a statistical power of 90% to detect a genetic OR of 1.3, assuming an allelic frequency of 10%, considering an unpaired control 1:1 of the genetic factor.
  A prevalence of 10% of the disease in the target population was considered, an alpha significance level of 5%, bilateral hypothesis test.
Sampling Method: Probability Sample
Enrollment: 3974 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Population attributable risk fraction measured for the Polygenic Risk Score. Scale will range from 0 to maximum number of risk alleles. The higher the score, the higher the number of risk alleles (worse). | through study completion, an average of 1 year
  Population attributable risk fraction of atherosclerotic cardiovascular diseases adjusted for other risk factors related to: diet, physical exercise, smoking, alcoholism, chronic disease history (diabetes, hypertension, dyslipidemia, etc) and biochemical parameters.
Polymorphisms genes as an independent risk factor for the occurrence of Acute Myocardial infarction (AMI), stroke and peripherical arterial thrombotic-ischemic events | through study completion, an average of 1 year
  As it is a case-control study, there will be no follow-up for the occurrence of clinical events. Therefore, we will assess exposures to traditional risk factors to cardiovascular events (MI, Stroke and acute peripheral atherothrombotic event) in combination with genomic data (polygenic risk score) in both cases and controls, and these exposures will be expressed as odds ratios. Multiple logistic regression models will be built to adjust and determine the strengths of association between demographic variables, traditional risk factors and genetic data

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Avezum, MD, PhD, Study Chair — Hospital Alemão Oswaldo Cruz
Locations (41):
- Brazil (41):
  - Acurácia Serviços Médicos, Rio Branco, Acre
  - Centro de Pesquisas Clínicas Dr. Marco Mota HCOR, Maceió, Alagoas
  - Centro de Pesquisa Clínica do Coração, Aracaju, Ceará
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Hospital Evangélico de Vila Velha, Vila Velha, Espírito Santo
  - Hospital Universitário Cassiano Antônio de Moraes, Vitória, Espírito Santo
  - Hospital e Clínica São Roque, Ipiaú, Estado de Bahia
  - Instituto Cárdio Pulmonar da Bahia, Salvador, Estado de Bahia
  - Universidade Federal de Goiás - UFG, Goiânia, Goiás
  - Hospital Universitário da Universidade Federal do Maranhão/HU/UFMA, São Luís, Maranhão
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande, Mato Grosso do Sul
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas da Universidade Federal do Triângulo Mineiro, Uberaba, Minas Gerais
  - Hospital Geral Filantrópico Universitário - Assoc. de Proteção à Maternidade e Infância de Cuiabá, Cuiabá, Mount
  - Hospital e Maternidade Angelina Caron, Campina Grande do Sul, Paraná
  - Núcleo de Pesquisa Clínica S/S, Curitiba, Paraná
  - Real Hospital Português de Beneficência em Pernambuco, Recife, Pernambuco
  - Hospital Universitário da Universidade Federal do Piauí, Teresina, Piauí
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Associação Dr. Bartholomeu Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Santa Casa de Misericórdia de Pelotas, Pelotas, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora Da Conceicao Sa, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Universitário de Santa Maria, Santa Maria, Rio Grande do Sul
  - Maestri e Kormann Consultoria Medico Cientifica, Blumenau, Santa Catarina
  - H&W Cardiologia LTDA, Joinville, Santa Catarina
  - Hospital Cirurgia, Aracaju, Sergipe
  - Hospital Municipal de Barueri, Barueri, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Scentryfar Pesquisa Clínica, Campinas, São Paulo
  - Hospital Carlos Fenando Malzoni, Matão, São Paulo
  - Braile Hospital Dia Ltda, São José do Rio Preto, São Paulo
  - Fundação Faculdade de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Instituto de Cardiologia HCFMUSP, São Paulo, São Paulo
  - Instituto de Pesquisa GNDI, São Paulo, São Paulo
  - Hospital Santa Paula, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Donnell MJ, Chin SL, Rangarajan S, Xavier D, Liu L, Zhang H, Rao-Melacini P, Zhang X, Pais P, Agapay S, Lopez-Jaramillo P, Damasceno A, Langhorne P, McQueen MJ, Rosengren A, Dehghan M, Hankey GJ, Dans AL, Elsayed A, Avezum A, Mondo C, Diener HC, Ryglewicz D, Czlonkowska A, Pogosova N, Weimar C, Iqbal R, Diaz R, Yusoff K, Yusufali A, Oguz A, Wang X, Penaherrera E, Lanas F, Ogah OS, Ogunniyi A, Iversen HK, Malaga G, Rumboldt Z, Oveisgharan S, Al Hussain F, Magazi D, Nilanont Y, Ferguson J, Pare G, Yusuf S; INTERSTROKE investigators. Global and regional effects of potentially modifiable risk factors associated with acute stroke in 32 countries (INTERSTROKE): a case-control study. Lancet. 2016 Aug 20;388(10046):761-75. doi: 10.1016/S0140-6736(16)30506-2. Epub 2016 Jul 16. PMID 27431356
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Stram DO. Design, Analysis, and Interpretation of Genome-Wide Association Scans. Springer; 2014.
- [Background] Gauderman WJ MJ. Quanto 1.1: A computer program for power and sample size calculations for genetic-epidemiology studies. 2006.
- [Background] Yusuf S, Joseph P, Rangarajan S, Islam S, Mente A, Hystad P, Brauer M, Kutty VR, Gupta R, Wielgosz A, AlHabib KF, Dans A, Lopez-Jaramillo P, Avezum A, Lanas F, Oguz A, Kruger IM, Diaz R, Yusoff K, Mony P, Chifamba J, Yeates K, Kelishadi R, Yusufali A, Khatib R, Rahman O, Zatonska K, Iqbal R, Wei L, Bo H, Rosengren A, Kaur M, Mohan V, Lear SA, Teo KK, Leong D, O'Donnell M, McKee M, Dagenais G. Modifiable risk factors, cardiovascular disease, and mortality in 155 722 individuals from 21 high-income, middle-income, and low-income countries (PURE): a prospective cohort study. Lancet. 2020 Mar 7;395(10226):795-808. doi: 10.1016/S0140-6736(19)32008-2. Epub 2019 Sep 3. PMID 31492503
- [Background] Roberts R, Chang CC, Hadley T. Genetic Risk Stratification: A Paradigm Shift in Prevention of Coronary Artery Disease. JACC Basic Transl Sci. 2021 Mar 22;6(3):287-304. doi: 10.1016/j.jacbts.2020.09.004. eCollection 2021 Mar. PMID 33778213
- [Background] Lu H, Zhang J, Chen YE, Garcia-Barrio MT. Integration of Transformative Platforms for the Discovery of Causative Genes in Cardiovascular Diseases. Cardiovasc Drugs Ther. 2021 Jun;35(3):637-654. doi: 10.1007/s10557-021-07175-1. Epub 2021 Apr 15. PMID 33856594
- [Background] Vrablik M, Dlouha D, Todorovova V, Stefler D, Hubacek JA. Genetics of Cardiovascular Disease: How Far Are We from Personalized CVD Risk Prediction and Management? Int J Mol Sci. 2021 Apr 17;22(8):4182. doi: 10.3390/ijms22084182. PMID 33920733
- [Background] Lanas F, Seron P, Lanas A. Coronary heart disease and risk factors in latin america. Glob Heart. 2013 Dec;8(4):341-8. doi: 10.1016/j.gheart.2013.11.005. PMID 25690636
- [Background] Piegas LS, Avezum A, Pereira JC, Neto JM, Hoepfner C, Farran JA, Ramos RF, Timerman A, Esteves JP; AFIRMAR Study Investigators. Risk factors for myocardial infarction in Brazil. Am Heart J. 2003 Aug;146(2):331-8. doi: 10.1016/S0002-8703(03)00181-9. PMID 12891204
- [Background] Teo KK, Ounpuu S, Hawken S, Pandey MR, Valentin V, Hunt D, Diaz R, Rashed W, Freeman R, Jiang L, Zhang X, Yusuf S; INTERHEART Study Investigators. Tobacco use and risk of myocardial infarction in 52 countries in the INTERHEART study: a case-control study. Lancet. 2006 Aug 19;368(9536):647-58. doi: 10.1016/S0140-6736(06)69249-0. PMID 16920470
- [Background] Gerstein HC, Islam S, Anand S, Almahmeed W, Damasceno A, Dans A, Lang CC, Luna MA, McQueen M, Rangarajan S, Rosengren A, Wang X, Yusuf S. Dysglycaemia and the risk of acute myocardial infarction in multiple ethnic groups: an analysis of 15,780 patients from the INTERHEART study. Diabetologia. 2010 Dec;53(12):2509-17. doi: 10.1007/s00125-010-1871-0. Epub 2010 Aug 14. PMID 20711717
- [Background] Schmidt MI, Duncan BB, Azevedo e Silva G, Menezes AM, Monteiro CA, Barreto SM, Chor D, Menezes PR. Chronic non-communicable diseases in Brazil: burden and current challenges. Lancet. 2011 Jun 4;377(9781):1949-61. doi: 10.1016/S0140-6736(11)60135-9. Epub 2011 May 9. PMID 21561658
- [Background] Pinho Nde A, Pierin AM. Hypertension control in brazilian publications. Arq Bras Cardiol. 2013 Sep;101(3):e65-73. doi: 10.5935/abc.20130173. PMID 24061761
- [Background] Walldius G, Jungner I, Holme I, Aastveit AH, Kolar W, Steiner E. High apolipoprotein B, low apolipoprotein A-I, and improvement in the prediction of fatal myocardial infarction (AMORIS study): a prospective study. Lancet. 2001 Dec 15;358(9298):2026-33. doi: 10.1016/S0140-6736(01)07098-2. PMID 11755609
- [Background] Iqbal R, Anand S, Ounpuu S, Islam S, Zhang X, Rangarajan S, Chifamba J, Al-Hinai A, Keltai M, Yusuf S; INTERHEART Study Investigators. Dietary patterns and the risk of acute myocardial infarction in 52 countries: results of the INTERHEART study. Circulation. 2008 Nov 4;118(19):1929-37. doi: 10.1161/CIRCULATIONAHA.107.738716. Epub 2008 Oct 20. PMID 18936332
- [Background] Leon DA, Saburova L, Tomkins S, Andreev E, Kiryanov N, McKee M, Shkolnikov VM. Hazardous alcohol drinking and premature mortality in Russia: a population based case-control study. Lancet. 2007 Jun 16;369(9578):2001-2009. doi: 10.1016/S0140-6736(07)60941-6. PMID 17574092
- [Background] Leong DP, Smyth A, Teo KK, McKee M, Rangarajan S, Pais P, Liu L, Anand SS, Yusuf S; INTERHEART Investigators. Patterns of alcohol consumption and myocardial infarction risk: observations from 52 countries in the INTERHEART case-control study. Circulation. 2014 Jul 29;130(5):390-8. doi: 10.1161/CIRCULATIONAHA.113.007627. Epub 2014 Jun 13. PMID 24928682
- [Background] Rosengren A, Hawken S, Ounpuu S, Sliwa K, Zubaid M, Almahmeed WA, Blackett KN, Sitthi-amorn C, Sato H, Yusuf S; INTERHEART investigators. Association of psychosocial risk factors with risk of acute myocardial infarction in 11119 cases and 13648 controls from 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):953-62. doi: 10.1016/S0140-6736(04)17019-0. PMID 15364186
- [Background] Gladding PA, Legget M, Fatkin D, Larsen P, Doughty R. Polygenic Risk Scores in Coronary Artery Disease and Atrial Fibrillation. Heart Lung Circ. 2020 Apr;29(4):634-640. doi: 10.1016/j.hlc.2019.12.004. Epub 2019 Dec 27. PMID 31974023
- [Background] van Rheenen W, Peyrot WJ, Schork AJ, Lee SH, Wray NR. Genetic correlations of polygenic disease traits: from theory to practice. Nat Rev Genet. 2019 Oct;20(10):567-581. doi: 10.1038/s41576-019-0137-z. PMID 31171865
- [Background] Li R, Chen Y, Ritchie MD, Moore JH. Electronic health records and polygenic risk scores for predicting disease risk. Nat Rev Genet. 2020 Aug;21(8):493-502. doi: 10.1038/s41576-020-0224-1. Epub 2020 Mar 31. PMID 32235907
- [Background] Anand SS, Xie C, Pare G, Montpetit A, Rangarajan S, McQueen MJ, Cordell HJ, Keavney B, Yusuf S, Hudson TJ, Engert JC; INTERHEART Investigators. Genetic variants associated with myocardial infarction risk factors in over 8000 individuals from five ethnic groups: The INTERHEART Genetics Study. Circ Cardiovasc Genet. 2009 Feb;2(1):16-25. doi: 10.1161/CIRCGENETICS.108.813709. Epub 2009 Jan 23. PMID 20031563
- [Background] Moura RR, Coelho AV, Balbino Vde Q, Crovella S, Brandao LA. Meta-analysis of Brazilian genetic admixture and comparison with other Latin America countries. Am J Hum Biol. 2015 Sep-Oct;27(5):674-80. doi: 10.1002/ajhb.22714. Epub 2015 Mar 26. PMID 25820814
- [Background] Pena SDJ, Santos FR, Tarazona-Santos E. Genetic admixture in Brazil. Am J Med Genet C Semin Med Genet. 2020 Dec;184(4):928-938. doi: 10.1002/ajmg.c.31853. Epub 2020 Nov 18. PMID 33205899
- [Background] Kehdy FS, Gouveia MH, Machado M, Magalhaes WC, Horimoto AR, Horta BL, Moreira RG, Leal TP, Scliar MO, Soares-Souza GB, Rodrigues-Soares F, Araujo GS, Zamudio R, Sant Anna HP, Santos HC, Duarte NE, Fiaccone RL, Figueiredo CA, Silva TM, Costa GN, Beleza S, Berg DE, Cabrera L, Debortoli G, Duarte D, Ghirotto S, Gilman RH, Goncalves VF, Marrero AR, Muniz YC, Weissensteiner H, Yeager M, Rodrigues LC, Barreto ML, Lima-Costa MF, Pereira AC, Rodrigues MR, Tarazona-Santos E; Brazilian EPIGEN Project Consortium. Origin and dynamics of admixture in Brazilians and its effect on the pattern of deleterious mutations. Proc Natl Acad Sci U S A. 2015 Jul 14;112(28):8696-701. doi: 10.1073/pnas.1504447112. Epub 2015 Jun 29. PMID 26124090
- [Background] Carneiro-Proietti ABF, Kelly S, Miranda Teixeira C, Sabino EC, Alencar CS, Capuani L, Salomon Silva TP, Araujo A, Loureiro P, Maximo C, Lobo C, Flor-Park MV, Rodrigues DOW, Mota RA, Goncalez TT, Hoppe C, Ferreira JE, Ozahata M, Page GP, Guo Y, Preiss LR, Brambilla D, Busch MP, Custer B; International Component of the NHLBI Recipient Epidemiology and Donor Evaluation Study (REDS-III). Clinical and genetic ancestry profile of a large multi-centre sickle cell disease cohort in Brazil. Br J Haematol. 2018 Sep;182(6):895-908. doi: 10.1111/bjh.15462. Epub 2018 Jul 19. PMID 30027669
- [Background] Cubillos-Angulo JM, Arriaga MB, Melo MGM, Silva EC, Alvarado-Arnez LE, de Almeida AS, Moraes MO, Moreira ASR, Lapa E Silva JR, Fukutani KF, Sterling TR, Hawn TR, Kritski AL, Oliveira MM, Andrade BB. Polymorphisms in interferon pathway genes and risk of Mycobacterium tuberculosis infection in contacts of tuberculosis cases in Brazil. Int J Infect Dis. 2020 Mar;92:21-28. doi: 10.1016/j.ijid.2019.12.013. Epub 2019 Dec 13. PMID 31843671
- [Background] Kim V, Wal TV, Nishi MY, Montenegro LR, Carrilho FJ, Hoshida Y, Ono SK. Brazilian cohort and genes encoding for drug-metabolizing enzymes and drug transporters. Pharmacogenomics. 2020 Jun;21(9):575-586. doi: 10.2217/pgs-2020-0013. Epub 2020 Jun 3. PMID 32486903
- [Background] Colares VS, Titan SM, Pereira Ada C, Malafronte P, Cardena MM, Santos S, Santos PC, Fridman C, Barros RT, Woronik V. MYH9 and APOL1 gene polymorphisms and the risk of CKD in patients with lupus nephritis from an admixture population. PLoS One. 2014 Mar 21;9(3):e87716. doi: 10.1371/journal.pone.0087716. eCollection 2014. PMID 24658608
- [Derived] Alves de Oliveira H Junior, de Menezes Neves PDM, de Figueiredo Oliveira GB, Moreira FR, Pintao MCT, Rocha VZ, de Souza Rocha C, Katz VN, Ferreira EN, Rojas-Malaga D, Viana CF, da Silva FF, Vidotti JJ, Felicio NM, de Araujo Vitor L, Cesar KG, Araujo da Silva C, de Oliveira Alves LB, Avezum A. Impact of genetic background as a risk factor for atherosclerotic cardiovascular disease: A protocol for a nationwide genetic case-control (CV-GENES) study in Brazil. PLoS One. 2024 Mar 13;19(3):e0289439. doi: 10.1371/journal.pone.0289439. eCollection 2024. PMID 38478535